CLINICAL TRIAL: NCT00263289
Title: The Effect of Preprocedural Fasting on Vomiting Frequency in Children Administered Nitrous Oxide -Oxygen Inhalation Analgesia for Dental Treatment
Brief Title: Preprocedural Fasting and Nitrous Oxide -Oxygen Inhalation Analgesia for Dental Treatment of Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: n20kup-HMO-CTIL
Record Dates: First submitted 2005-12-07; First posted 2005-12-08 (Estimated); Last update posted 2005-12-08 (Estimated); Status verified 2005-12

CONDITIONS: Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Time Perspective: Other

INTERVENTIONS:
Procedure: preprocedural fasting

SUMMARY:
Nitrous oxide analgesia is used routinely for the dental treatment of anxious or uncooperative pediatric patients. In many instances it is used alone without any supplemental oral premedication. A controversy exists among pediatric dentists and pediatric dental departments regarding the need to apply pre-procedural fasting (PF) or other limitations on children undergoing dental treatment with nitrous oxide alone.The purpose of this study is to investigate the association between PF and the frequency of vomiting in pediatric patients receiving dental treatment with nitrous oxide analgesia.

DETAILED DESCRIPTION:
Materials and methods The experimental protocol will be submitted for approved by the Institutional Human Subjects Ethics committee of Hadassah-Hebrew University School of Dental l Medicine. Informed consent will be obtained from all parents or legal guardians of participating subjects.

Subjects All pediatric patients attending the graduate student pediatric dental clinic of the Department of Pediatric Dentistry at Hadassah Clinic in need of at least two restorative treatment sessions with the use of nitrous oxide will be included. All participants must be in good health (ASA I). Prior to one session subjects will be restricted and have a preprocedural fasting as per the following guidelines: All subjects will be without solids (including milk) for at least 4 hours prior to nitrous oxide administration and without clear liquids 2 hours before treatment. On the alternative session subjects will have no restrictions on their food or liquid intake.

Evaluation

A survey will be given to parents prior to treatment and information regarding the following will be gathered:

Age, previous nitrous oxide experience, history of vomiting or nausea (motion sickness, foods etc), last mea: what and when? The resident administering treatment will record the following: Duration of inhalation administration, percentage of nitrous oxide and flow rate, steady or fluctuating, occurrence of vomiting during or immediately following treatment.

Statistical analysis of data will determine the incidence of vomiting and if any significant differences between the two sessions exist.

ELIGIBILITY:
Inclusion Criteria:

- All pediatric patients attending the graduate student pediatric dental clinic of the Department of Pediatric Dentistry at Hadassah Clinic in need of at least two restorative treatment sessions with the use of nitrous oxide will be included. All participants must be in good health (ASA I).

Exclusion Criteria:

-

Ages: 4 Years to 17 Years | Sex: All
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Ari Kupietzky, DMD MSc, Principal Investigator — Clinical Instructor, Department of Pediatric Dentistry, Hadassah School of Dental Medicine
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel